CLINICAL TRIAL: NCT02373618
Title: Dry Needling Versus Conventional Physical Therapy in Patients With Plantar Fasciitis: a Multi-center Randomized Clinical Trial
Brief Title: Dry Needling Versus Conventional Physical Therapy in Patients With Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, DPT FAAOMPT, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT0002
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2016-07

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: DN and Conventional PT (Experimental)
  Interventions: Other: DN and conventional PT
- Active Comparator: Conventional PT (Active Comparator)
  Interventions: Other: Conventional PT

INTERVENTIONS:
Other: DN and conventional PT — Dry needling to the foot and lower leg. Up to 8 sessions over 4 weeks. Also conventional PT including: ultrasound, stretching, strengthening, cryotherapy and manual therapy to the foot and lower leg.
  Arms: Experimental: DN and Conventional PT
Other: Conventional PT — Conventional physical therapy includes ultrasound, strengthening, cryotherapy, and manual therapy up to 8 sessions over 4 weeks.
  Arms: Active Comparator: Conventional PT

SUMMARY:
The purpose of this research is to compare patient outcomes following treatment of plantar fasciitis with conventional physical therapy (stretching, strengthening, ultrasound, manual therapy, and cryotherapy) and conventional physical therapy plus dry needling. Physical therapists commonly use conventional physical therapy techniques and dry needling to treat plantar fasciitis, and this study is attempting to find out if the addition of dry needling to conventional physical therapy is more effective than conventional physical therapy alone.

DETAILED DESCRIPTION:
Patients with plantar fasciitis will be randomly assigned to receive 1-2 treatments per week for 4 weeks of either: (1) Dry Needling and conventional physical therapy, or the (2) Conventional physical therapy (stretching, strengthening, ultrasound, manual therapy, and cryotherapy)

ELIGIBILITY:
Inclusion Criteria:

1. Report of at least 3 months of heel pain
2. Patient has not had physical therapy, massage therapy, chiropractic treatment, or injections for plantar heel pain in the least 4 weeks.
3. Diagnosis of plantar heel pain with ALL of the following positive clinical signs:

   * "First---step" pain upon weight bearing in the morning OR after sitting for a period of time
   * Pain localized over the medial calcaneal tubercle
   * Increased pain with extended walking OR standing >15 minutes
4. Plantar heel pain greater than or equal to 2/10 (NPRS 0-10 Scale)

Exclusion Criteria:

1. Report of red flags to manual physical therapy to include: hypertension, infection, diabetes, peripheral neuropathy, heart disease, stroke, chronic ischemia, edema, severe varicosities, tumor, metabolic disease, prolonged steroid use, fracture, RA, osteoporosis, severe vascular disease, malignancy, etc.
2. History of previous surgery to the tibia, fibula, ankle joint, or foot.
3. History of arthrosis or arthritis of the ankle and/or foot.
4. History of significant ankle and/or foot instability.
5. Two or more positive neurologic signs consistent with nerve root compression, including any two of the following:

   * Muscle weakness involving a major lower extremity muscle group
   * Diminished lower extremity patella or Achilles tendon reflexes
   * Diminished / absent sensation in any lower extremity dermatome
6. Involvement in litigation or worker's compensation regarding their foot pain.
7. Any condition that might contraindicate the use of electro---needling
8. The patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Change in Lower Extremity Functional Scale | Baseline, 1 week, 4 weeks, 3 months
  20 questions each worth 0-4 points with maximum score of 80 points possible. Do not convert to a 20 questions, each worth 0-4 points with maximum score of 80 points possible
Change in First Step Pain in the Morning (NPRS) | Baseline, 1 week, 4 weeks, 3 months
Change in Activity Pain (NPRS) | Baseline, 1 week, 4 weeks, 3 months
  Average pain level during standing and walking.
Change in Pain Intensity (NPRS) | Baseline, 1 week, 4 weeks, 3 months
Change in Foot Functional Index Pain | Baseline, 1 week, 4 weeks, 3 months
  5 questions each worth 0-10 points with maximum score of 50 points possible.
Change in Foot Functional Index Disability | Baseline, 1 week, 4 weeks, 3 months
  9 questions each worth 0-10 points with maximum score of 90 points possible
Change in Foot Functional Index Activity Limitation | Baseline, 1 week, 4 weeks, 3 months
  3 questions each worth 0-10 points with maximum score of 30 points possible
Change in Foot Functional Index Total | Baseline, 1 week, 4 weeks, 3 months
  3 questions each worth 0-10 points with maximum score of 30 points possible

SECONDARY OUTCOMES:
Change in Global Rating of Change Score | 1 week, 4 weeks, 3 months
Change in Medicine Intake (Frequency of pain medication) | Baseline, 3 months
  Frequency of pain medication, including over-the-counter or narcotics for plantar fasciitis

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT FAAOMPT, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Alabama Physical Therapy & Acupuncture, Montgomery, Alabama, United States